CLINICAL TRIAL: NCT06626438
Title: Treatable Traits in Interstitial Lung Disease
Acronym: TTRILD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Western Australia (Other)
Collaborators: Fiona Stanley Hospital (Other); Sir Charles Gairdner Hospital (Other)
Responsible Party: Principal Investigator, Megan Harrison, Dr., The University of Western Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGS0000006668; MRFF2022914 (Other Grant/Funding Number: Medical Research Future Fund (Australian Government Department of Health and Aging))
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Interstitial Lung Diseases (ILD)
Keywords: treatable traits; interstitial lung disease; pulmonary fibrosis; multidisciplinary
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatable Traits model of care (Experimental): Embedded multidisciplinary clinic. This involves multidimensional assessment of patients with MDT review to determine presence of treatable traits and their specific management.
  Interventions: Other: Treatable traits model of care
- Standard of Care (No Intervention): Standard of care where physician-led ILD clinic. All referrals and comorbidity management as guided by physician.

INTERVENTIONS:
Other: Treatable traits model of care — Embedded multidisciplinary clinic with treatable traits model of care.
  Arms: Treatable Traits model of care

SUMMARY:
The goal of this clinical trial is to learn if a personalised treatment model of care "treatable traits" can improve quality of life and disease progression in patients with interstitial lung disease.

The main question it aims to answer is, will providing a treatable traits model of care improve health-related quality of life (HRQoL) (primary outcome), symptoms, anxiety, physical activity, and body composition (secondary outcomes).

Researchers will compare the treatable traits model to standard of care.

Participants in both arms will complete surveys, a Dual-Energy X-Ray Absorptiometry (DEXA) and whole-body composition scan, lung function and blood tests. Those in the intervention (TT) arm will be seen in a multidisciplinary clinic where they are seen by an ILD doctor, physiotherapist, psychologist, and dietitian.

DETAILED DESCRIPTION:
RCT to compare treatable traits (TT) model of care to standard practice. Primary endpoints reviewed will be health-related QOL as defined by the validated King's Brief Interstitial Lung Disease (KB-ILD) questionnaire. Secondary endpoints will include progression free survival (the time to disease progression or death from any cause), all-cause hospitalisation and mortality, and economic evaluation (comparison of per person direct and indirect costs intervention vs standard of care).

Patients included will be those over 18yo with an interstitial lung disease across hospitals in Western Australia. Target study number will be 55 per arm. Participants will be randomised via an online randomisation system (REDCAP) in a 1:1 fashion to standard or care of the TT MDT clinic. Randomisation will be stratified with a 50% IPF limit and according to severity (mild, moderate and severe from FVC). Participants and clinicians will not be blinded to group allocation. Statistician will be blinded for data analysis.

The embedded clinic will involve multidimensional assessment of patients. At the clinic, the patient will be assessed by a nurse, physiotherapist, psychologist, dietician, and physician. At the end of the clinic the team will meet to discuss each patient and devise a plan to optimise the management of TTs for that individual.

Multidimensional assessment will include demographics, co-morbidities, medications, exposures, blood results, prior investigations, and MDT diagnosis. Questionnaires completed at time of enrolment include KB-ILD (assess QOL), SF26 QOL), Leister Cough questionnaire (Cough), Stop-bang (OSA), mMRC (SOB), fatigue severity score (Fatigue), PGSGASF (nutritional status), perceived stress score (anxiety), GAD score (anxiety), PHQ9 (depression).

Other assessments include lung function, blood testing, sputum assessment, HRCT. Physiotherapy assessments will include 1 minute STS, 6MWT, DEXA scan. Nutritional assessment will be based on BMI and PG-SGA scores.

Interventions provided include standard of care medications (anti-fibrotic and immunosuppressive therapies as per guidelines). Specific physiotherapy intervention will be pulmonary rehabilitation; dietician input will involve dietary counselling and consideration of oral nutritional supplements. Psychology intervention will be self-management strategies or referral to individual psychology.

ELIGIBILITY:
Inclusion Criteria: Patients with a new or pre-existing diagnosis of fibrotic ILD who receive care via the Fiona Stanley Hospital (FSH) or Sir Charles Gairdner Hospital (SCGH) ILD service will be invited to participate. This ILD diagnosis must be made through an ILD MDT.

Included participants will be aged ≥ 18 years with a physician-confirmed diagnosis of fibrotic ILD. Fibrotic ILD is defined as presence of fibrotic changes on CT in the opinion of the investigator. All ILD subtypes, excluding sarcoidosis, will be included. Participants will need to be able to provide consent to participate and be established on stable ILD treatment for 1 month prior to study initiation.

Exclusion Criteria: Participants will be excluded if they have experienced an acute exacerbation 4 weeks prior to starting the study or are expected to experience either a transplant or death during the study period. Active suicidality, severe depression, active psychosis or mania, or other severe psychiatric concerns that require more intensive treatment. Any such participants could be referred for individual therapy and/or psychiatric treatment that would be more appropriate for their needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | from enrolment to 6 months post intervention.
  Kings brief interstitial lung disease score that has been validated in quality of life for ILD patients.

SECONDARY OUTCOMES:
Progression free survival | from enrolment to 12 months post intervention (14 months post enrolment)
  the time to disease progression or death from any cause.
Exercise capacity | from enrolment to 12 months post intervention (14 months post enrolment)
  6 minute walk test assessment

OTHER OUTCOMES:
Economic evaluation | from enrolment to 12 months post intervention (14 months post enrolment)
  * A comparison of per person direct (health system and all patient expenses) and indirect (lost productivity) costs will be performed for the treatable trait program versus standard care.
  * Direct costs will include: staff time; visits to the GP, specialist or emergency room; hospitalisation; and use of chronic disease services including pulmonary rehabilitation, nursing and allied health services.
  * Patient expenses include transportation and parking costs, co-payments for medications and consultations, and costs of equipment and household adaptations

CONTACTS AND LOCATIONS:
Overall Officials: Yuben Moodley, MBSS, FRACP, MD, PHD, Principal Investigator — The University of Western Australia
Locations (2):
- Australia (2):
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT06626438/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT06626438/ICF_001.pdf